CLINICAL TRIAL: NCT00234780
Title: In Home Hospital Care Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6427; MCHB MCJ-360831; NINR 5 R01NR04501-03
Record Dates: First submitted 2005-10-05; First posted 2005-10-07 (Estimated); Last update posted 2007-08-16 (Estimated); Status verified 2005-10

CONDITIONS: Common Acute Problems
Keywords: acute home care

INTERVENTIONS:
Procedure: pediatric nursing used in home to avoid hospitalization

SUMMARY:
To assess the hypothesis that In Home Hospital Care (IHHC) is as safe and effective, less burdensome to families, and less expensive for care of common acute pediatric problems now managed with hospitalization.

DETAILED DESCRIPTION:
A randomized trial compared health care systems with and without IHHC. Eligible children presented to the Emergency Department of our medical center, had common acute problems, and were considered for hospital admission.

Physicians decided disposition from the emergency department. Note that subjects were not randomized directly to IHHC but to a system of care that either included IHHC or did not. To allow best use of scarce home nursing resources, we used a disproportionate selection favoring the system with IHHC.

Quality measures included adverse events, parent anxiety and satisfaction with care, family disruption, and perceived child health.

ELIGIBILITY:
Inclusion Criteria:

Randomized from acute care clients presenting in Emergency Department to IHHC

Exclusion Criteria:

Randomized from acute care clients presenting in Emergency Department to inpatient hospital care.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200
Dates: Start 1997-10; Study Completion 2000-08

PRIMARY OUTCOMES:
IHHC delivers a more valuable service at lower cost.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth M. McConnochie, MD,MPH, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States